CLINICAL TRIAL: NCT01894984
Title: Clinical Observation of the Efficacy and Safety of Risperidone Long-Acting Injection (Risperdal Consta) in the Treatment of Schizophrenia in China
Brief Title: An Observational Study to Evaluate Efficacy and Safety of Risperidone Long-Acting Injection for Treatment of Schizophrenia
Status: Terminated | Type: Observational
Why Stopped: The study was terminated because of high dropout rate.
Sponsor: Xian-Janssen Pharmaceutical Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR013483; RISSCH4191
Record Dates: First submitted 2013-07-03; First posted 2013-07-10 (Estimated); Results first posted 2013-11-08 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-04

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Risperidone; Risperdal Consta; Oral antipsychotic
MeSH Terms: conditions — Schizophrenia | interventions — Risperidone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Risperidone: Risperidone will be administered as intramuscular injection at a starting dose of either 25 milligram (mg) or 37.5 mg or 50 mg (starting dose will be decided on the basis of the disease severity), every two weeks, up to Week 24, wherein after Week 8, dose may be increased or decreased at physician discretion. For first three weeks, previous oral antipsychotic drug (Benzodiazepines or Selective serotonin reuptake inhibitor [SSRI]) will be maintained and will cease at Week 3.
  Interventions: Drug: Risperidone
- Oral atypical anti-psychotic: Oral atypical anti-psychotic for example, olanzapine, risperidone, quetiapine etc will be administered as per Investigator's discretion.
  Interventions: Drug: Oral atypical anti-psychotic

INTERVENTIONS:
Drug: Risperidone — This is an observational study. Risperidone will be administered as intramuscular injection at a starting dose of either 25 milligram (mg) or 37.5 mg or 50 mg (starting dose will be decided on the basis of the disease severity), every two weeks, up to Week 24, wherein after Week 8, dose may be increased or decreased at physician discretion. For first three weeks, previous oral antipsychotic drug (Benzodiazepines or Selective serotonin reuptake inhibitor [SSRI]) will be maintained and will cease at Week 3.
  Other Names: Risperdal Consta
  Groups: Risperidone
Drug: Oral atypical anti-psychotic — This is an observational study. Oral atypical anti-psychotic for example, olanzapine, risperidone, quetiapine etc will be administered as per Investigator's discretion.
  Groups: Oral atypical anti-psychotic

SUMMARY:
The purpose of this study is to evaluate the long-term treatment efficacy, and safety of risperidone long-acting injection in participants with schizophrenia (psychiatric disorder with symptoms of emotional instability, detachment from reality, often with delusions and hallucinations, and withdrawal into the self).

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), multi-center (conducted in more than one center), prospective (study following participants forward in time) and observational study of risperidone long-acting injection in participants with schizophrenia. The study consists of 2 parts: Screening (that is, 28 days before study commences on Day 1) and Treatment (that is, Week 1-24). All the eligible participants (after risperidone intolerance test during screening) will be receiving risperidone as intramuscular injection (injection of a substance into a muscle) at a dose of, either 25 milligram (mg), 37.5 mg or 50 mg every two weeks. Efficacy of the participants will be primarily evaluated through Positive and Negative Syndrome Scale. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18-65 years
* Participant must meet the diagnostic criteria for schizophrenia or schizophreniform disorder according to Diagnostic and Statistical Manual of Mental Disorders, fourth edition (DSM-IV)-TM
* Total course of disease no more than 5 years
* According to physician's discretion, participants need to be changed to risperidone long-acting injection and other atypical anti-psychotic drug
* Participant or their legally acceptable representatives must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study

Exclusion Criteria:

* Significant risk of suicidal or violent behavior, as clinically assessed by the Investigator
* Have aggressive behavior and excited , restless
* History or current symptoms of tardive dyskinesia; neuroleptic malignant syndrome; evidence of dysfunction of liver and kidney and other severe physical diseases; and severe, life-threatening allergic reaction to any drug
* Known hypersensitivity to risperidone
* Female participant who is pregnant or breastfeeding or planning to become pregnant during the study period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participant must meet the diagnostic criteria for schizophrenia or schizophreniform disorder according to Diagnostic and Statistical Manual of Mental Disorders, fourth edition (DSM-IV)
Sampling Method: Non-Probability Sample
Enrollment: 640 (Actual)
Dates: Start 2007-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xian-Janssen Pharmaceutical Ltd., China Clinical Trial, Study Director — Xian-Janssen Pharmaceutical Ltd.

RESULTS

PARTICIPANT FLOW:
Groups:
- Risperidone: Risperidone was administered as intramuscular injection at a starting dose of either 25 milligram (mg) or 37.5 mg or 50 mg (starting dose was decided on the basis of the disease severity), every two weeks, up to Week 24, wherein after Week 8, dose may had been increased or decreased at Investigator's discretion. For first three weeks, previous oral antipsychotic drug (benzodiazepines or selective serotonin reuptake inhibitor [SSRI]) was maintained and ceased at Week 3.
- Oral Atypical Anti-psychotic: Oral atypical anti-psychotic for example, olanzapine, risperidone, quetiapine etc was administered as per Investigator's discretion.
Period: Overall Study
Arm/Group | Risperidone | Oral Atypical Anti-psychotic
Started | 396 | 244
Completed | 82 | 69
Not Completed | 314 | 175
Not completed — Other | 314 | 175

BASELINE CHARACTERISTICS:
Population: "N" (number of participants analyzed) signifies the participants evaluable for this measure.
Groups:
- Total: Total of all reporting groups
Arm/Group | Risperidone | Oral Atypical Anti-psychotic | Total
Number analyzed (Participants) | 396 | 243 | 639
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age is provided for 395 participants in Risperidone treatment group because complete date of birth detail is not available for one participant.
  Years | 27.4 (9.44) | 32.2 (11.62) | 29.2 (10.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 190 | 136 | 326
  Male | 206 | 107 | 313

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score at Week 24
Description: The PANSS is a 30-item scale designed to assess various symptoms of schizophrenia including delusions, grandiosity, blunted affect, poor attention, and poor impulse control. The 30 symptoms are rated on a 7-point scale that ranges from 1 (absent) to 7 (extreme psychopathology). The PANSS total score consists of the sum of all 30 PANSS items and ranges from 30 to 210. Higher scores indicate worsening.
Time Frame: Baseline and Week 24
Population: Intent to treat (ITT) population included all randomized participants who received at least one dose of study drug and had relevant efficacy evaluations.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Risperidone | Oral Atypical Anti-psychotic
Number analyzed (Participants) | 396 | 243
units on a scale
  Baseline | 74.7 (22.54) | 72.3 (20.49)
  Change at Week 24 | -36.5 (25.67) | -38.2 (24.06)

2. Secondary Outcome: Total Personal and Social Performance (PSP) Score
Description: The PSP is a clinician-rated scale that reflects social functioning in 4 domains of behavior (socially useful activities including work and study, personal and social relationships, self care, and disturbing and aggressive behaviors). The total score ranges from 1 to 100 (score of 71 to 100 will have a mild degree of difficulty; from 31 to 70, varying degrees of disability; less than or equal to 30, functioning so poorly as to require intensive supervision) divided into 10 equal intervals to rate the degree of difficulty (i=absent to vi=very severe) in each of the 4 domains.
Time Frame: Baseline and Week 24
Population: ITT population included all randomized participants who received at least one dose of study drug and had relevant efficacy evaluations.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Risperidone | Oral Atypical Anti-psychotic
Number analyzed (Participants) | 396 | 243
units on a scale
  Baseline | 52.1 (17.15) | 52.9 (16.00)
  Week 24 | 88.0 (10.25) | 82.3 (10.07)

3. Secondary Outcome: Clinical Global Impressions-Severity (CGI-S) Score
Description: The CGI-S rating scale is a 7-point global assessment that measures the clinician's impression of the severity of illness exhibited by a participant. A rating of 1 is equivalent to "Normal, not at all ill" and a rating of 7 is equivalent to "Among the most extremely ill participants". Higher scores indicate worsening.
Time Frame: Baseline and Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Risperidone | Oral Atypical Anti-psychotic
Number analyzed (Participants) | 396 | 243
units on a scale
  Baseline | 4.5 (1.15) | 4.6 (1.12)
  Week 24 | 1.5 (1.02) | 2.1 (1.14)

4. Secondary Outcome: Percentage of Participants With Relapse at Week 24
Description: Percentage of participants with relapse was assessed wherein relapse was defined as hospitalization due to the aggravation of psychiatric symptoms of disease condition.
Time Frame: Week 24
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Risperidone | Oral Atypical Anti-psychotic
Number analyzed (Participants) | 396 | 243
Percentage of Participants | 0.5 (22.54) | 1.6 (20.49)

5. Secondary Outcome: Percentage of Participants Attaining Remission Criteria
Description: Remission is defined as a clinical status where for each core symptoms (that are, delusions, conceptual disorganization, hallucinatory behavior, mannerisms and posturing unusual thought content, blunted affect, passive or apathetic social withdrawal and lack of spontaneity and flow of conversation) were assessed at a low-mild symptom intensity level, where such absent, borderline, or mild symptoms do not influence an individual's behavior.
Time Frame: Month 6
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Risperidone | Oral Atypical Anti-psychotic
Number analyzed (Participants) | 396 | 243
Percentage of Participants | 46 (22.54) | 68 (20.49)

6. Secondary Outcome: Number of Participants With Reasons for Discontinuation From Study Treatment
Description: Number of participants with reasons for discontinuation from study treatment is reported here because participants provided multiple reasons for discontinuation.
Time Frame: Month 6
Population: Analysis population included all enrolled participants.
Measure: Number; unit: Participants
Arm/Group | Risperidone | Oral Atypical Anti-psychotic
Number analyzed (Participants) | 396 | 244
Participants
  Physician Decision | 14 (22.54) | 11 (20.49)
  Adverse event | 24 | 3
  Lack of efficacy | 10 | 2
  Discontinuation from Treatment (more than 4 weeks) | 65 | 7
  Added other anti-psychotics | 10 | 3
  Change to other anti-psychotics | 57 | 18
  Lost to follow-up | 67 | 39
  Withdrawal by participant | 4 | 0
  Other (unspecified) | 128 | 106

ADVERSE EVENTS:
Time Frame: Baseline up to Week 24
Description: Safety population included all randomized participants who had at least baseline evaluations.
Arm/Group | Risperidone | Oral Atypical Anti-psychotic
Serious Adverse Events (participants affected / at risk) | 11/396 | 0/244
Other Adverse Events (participants affected / at risk) | 73/396 | 48/244
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Risperidone (N=396) | Oral Atypical Anti-psychotic (N=244)
Auditory hallucination (Psychiatric disorders) | 3 | 0
Headache (Nervous system disorders) | 1 | 0
Nervousness (Nervous system disorders) | 1 | 0
Schizophrenia (Psychiatric disorders) | 6 | 0
Persecutory delusion (Psychiatric disorders) | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Abnormal behaviour (Psychiatric disorders) | 1 | 0
Hallucination (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Risperidone (N=396) | Oral Atypical Anti-psychotic (N=244)
Hyperlipemia (Metabolism and nutrition disorders) | 0 | 3
Weight gain (Investigations) | 8 | 6
Extrapyramidal disease (Nervous system disorders) | 30 | 19
Anxiety (Psychiatric disorders) | 1 | 3
Schizophrenia (Psychiatric disorders) | 7 | 0
Akathisia (Psychiatric disorders) | 7 | 1
Somnolence (Psychiatric disorders) | 1 | 3
Amenorrhea (Reproductive system and breast disorders) | 11 | 1
Menstrual disorder (Reproductive system and breast disorders) | 8 | 2
Constipation (Gastrointestinal disorders) | 0 | 6
Hygrostomia (Gastrointestinal disorders) | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days